CLINICAL TRIAL: NCT02506205
Title: The Effect of LSVT LOUD for Mandarin-speaking Individuals With Hypokinetic Dysarthria Due to Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, National Taiwan University Hospital, National Taiwan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 201407035RINC
Record Dates: First submitted 2015-07-21; First posted 2015-07-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Hypokinetic Dysathria

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (1):
- LSVT LOUD (Experimental): LSVT LOUD was developed based on concepts of neuroplasticity, motor learning, skill acquisition and motor speech. LSVT LOUD trains laryngeal and respiratory functions through loud and effortful phonatory tasks (Ramig, Sapir, Countryman, Pawlas, O'Brien, Hoehn, & Thomson, 2001). It targets vocal intensity via stimulation of effortful speech productions with multiple repetitions and through encouraging self-calibrations of loud voice by patients. LSVT LOUD cues patients to speak loud (e.g., Fox et al., 2002; Ramig et al., 2001; Sapir et al., 2007). Having a single cue may increase treatment effects, as it reduces cognitive load in adults with PD because some of them develop cognitive deficits when PD progresses (Fox et al., 2002). Treatment is intensive, consisting of 4 individual sessions a week for 4 weeks, with 16 sessions in one month.
  Interventions: Behavioral: Lee Silverman Voice Treatment (SVLT) LOUD

INTERVENTIONS:
Behavioral: Lee Silverman Voice Treatment (SVLT) LOUD

SUMMARY:
A handful of studies have examined the effects of the Lee Silverman Voice Treatment (LSVT) LOUD on hypokinetic dysarthria in English speakers with Parkinson's disease (PD). Although LSVT LOUD has been found to be effective on improving these speaker's vocal intensity and increasing their speech intelligibility as well as speech function with Phase I evidence, no study has investigated whether Mandarin-speaking individuals with dysarthria secondary to PD would benefit from LSVT LOUD. In the proposed study, speech data of Mandarin-speaking individuals with hypokinetic dysarthria before and after speech therapy will be audio recorded and analyzed in order to examine the effects of LSVT LOUD on the speech function in this population. The same speech data will be played to Mandarin listeners in order to investigate the speech intelligibility of this population. It is hypothesized that Mandarin-speaking individuals with hypokinetic dysarthria secondary to PD will demonstrate reduced vocal intensity, reduced speech intelligibility and impaired speech function before they receive LSVT LOUD. They will improve these speech characteristics following speech therapy and will present with short-term maintenance effects.

ELIGIBILITY:
Inclusion Criteria:

1. Mandarin-speaking Taiwanese
2. Hypokinetic dysarthria due to Parkinson's disease
3. No other neurodegenerative diseases
4. No cognitive deficits
5. Age range 30 years and above

Exclusion Criteria:

1. Not able to follow verbal directions,
2. speech characteristics uncommon to Parkinson's disease

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Speech intelligibility | Immediate
  Speech intelligibility will be assessed by native Mandarin listeners' orthographic transcription accuracy and ratings based on a nine-point Likert scale (from 1 - very difficult to understand to 9 - very easy to understand).

SECONDARY OUTCOMES:
Speech function | Immdediate
  Speech function will be assessed using acoustic methods. E.g., vowel formant frequencies correlated with vowel articulation will be extracted and analyzed using Praat software.

OTHER OUTCOMES:
Quality of life measured by PDQ-39 | Immediate
  This area of assessment will be measured by Parkinson's Disease Questionnaire (PDQ-39) (Jenkinson, Fitzpatrick, Peto, Greenhall, & Hyman, 1997). This battery provides information on areas that affect participants' well-being and the degree affected.
Depression level measured by BDI-II | Immediate
  Some patients with PD develop depression that affects their daily life. Therefore, it is necessary to assess their depression level with Beck Depression Inventory-II (Beck, Steer, & Brown, 1996)
Cognitive status measured by MMSE | Immediate
  It is necessary to assess their cognitive status with Mini-mental State Examination (MMSE) (Folstein, Foistein, & McHugh, 1975) and the score will be used as the inclusion or exclusion criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Background] Darley FL, Aronson AE, Brown JR. Clusters of deviant speech dimensions in the dysarthrias. J Speech Hear Res. 1969 Sep;12(3):462-96. doi: 10.1044/jshr.1203.462. No abstract available. PMID 5811846
- [Background] Fox, C. M., Morrison, C. E., Ramig, L. O., & Sapir, S. (2002). Current perspectives on the Lee Silverman Voice Treatment (LSVT) for individuals with idiopathic Parkinson disease. American Journal of Speech-Language Pathology, 11: 111-123.
- [Background] Jeng JY, Weismer G, Kent RD. Production and perception of mandarin tone in adults with cerebral palsy. Clin Linguist Phon. 2006 Jan-Feb;20(1):67-87. doi: 10.1080/02699200400016539. PMID 16393799
- [Background] Liu, H.-M., Tseng, C.-H., & Tsao, F.-M. (2000). Perceptual and acoustic analysis of speech intelligibility in Mandarin-speaking young adults with cerebral palsy. Clinical Linguistics and Phonetics, 14: 447-464
- [Background] Ramig LO, Sapir S, Countryman S, Pawlas AA, O'Brien C, Hoehn M, Thompson LL. Intensive voice treatment (LSVT) for patients with Parkinson's disease: a 2 year follow up. J Neurol Neurosurg Psychiatry. 2001 Oct;71(4):493-8. doi: 10.1136/jnnp.71.4.493. PMID 11561033
- [Background] Sapir S, Spielman JL, Ramig LO, Story BH, Fox C. Effects of intensive voice treatment (the Lee Silverman Voice Treatment [LSVT]) on vowel articulation in dysarthric individuals with idiopathic Parkinson disease: acoustic and perceptual findings. J Speech Lang Hear Res. 2007 Aug;50(4):899-912. doi: 10.1044/1092-4388(2007/064). PMID 17675595
- [Background] Schulz GM, Grant MK. Effects of speech therapy and pharmacologic and surgical treatments on voice and speech in Parkinson's disease: a review of the literature. J Commun Disord. 2000 Jan-Feb;33(1):59-88. doi: 10.1016/s0021-9924(99)00025-8. PMID 10665513
- [Background] Whitehill TL, Wong LL. Effect of intensive voice treatment on tone-language speakers with Parkinson's disease. Clin Linguist Phon. 2007 Nov-Dec;21(11-12):919-25. doi: 10.1080/02699200701602045. PMID 17972188